CLINICAL TRIAL: NCT05902026
Title: Validity and Reliability of the BETY-Biopsychosocial Questionnaire (BETY-BQ) in Individuals With Temporomandibular Dysfunction-Related Headache.
Brief Title: The BETY-Biopsychosocial Questionnaire (BETY-BQ) in Individuals With Temporomandibular Dysfunction-Related Headache
Status: Enrolling by invitation | Type: Observational
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Aysenur Tuncer, Principle Investigator, Hasan Kalyoncu University
Other Study IDs: 2023-61
Record Dates: First submitted 2023-06-04; First posted 2023-06-13 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-12

CONDITIONS: Temporomandibular Disorders; Headache
Keywords: Temporomandibular disorders; Headache; Exercise Therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders; Headache

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates the validity and reliability of the BETY- Biopsychosocial Questionnaire (BETY-BQ) as a biopsychosocial assessment tool in individuals with temporomandibular dysfunction-related headaches.

DETAILED DESCRIPTION:
It is known that pain is a powerful motivational component and creates a complex experience that cannot be explained by illness, injury, or structural problems alone. It is emphasized that pain, including temporomandibular dysfunction-related pain, has a multifactorial structure and that chronic pain is affected by biological, psychological, and social factors. Biological and psychosocial factors contribute to the predisposition and triggering of temporomandibular dysfunction-related headache symptoms. As with many chronic pain conditions, recent research reinforces the biopsychosocial nature of joint painful temporomandibular dysfunction (myalgia and arthralgia) and their interconnections with general health. Psychological, social, and functional problems of individuals with TMJ dysfunction-related headaches should be considered together, and treatment targets should be determined accordingly. The biopsychosocial being of humans is the main reason for this approach. BETY- Biopsychosocial Questionnaire (BETY-BQ) originates from the Cognitive Exercise Therapy Approach (CETA), an innovative exercise approach that targets holistic treatment techniques per the biopsychosocial model. This approach contains concepts including function-oriented trunk stabilization exercises, pain management, mood management (dance therapy-authentic movement), and sexual knowledge management which are combined. It was first used in patients with ankylosing spondylitis, and it was observed that besides its positive effects on disease activity, and also provided positive changes in anti-inflammatory parameters. CETA has taken place in the literature as a biopsychosocial exercise model that can be applied safely in individuals with Multiple Sclerosis. Patients with rheumatism, who have participated in CETA training since 2004, described their recovery characteristics in 2013. The questionary was finalized in 2017 by applying this feedback to repetitive statistics and rheumatic patients who did not participate in the group. Validity and reliability studies of the developed scale were conducted in individuals diagnosed with Fibromyalgia, Rheumatoid Arthritis, Osteoarthritis, and chronic neck and low back pain.

The temporomandibular joint is a complex structure consisting of masticatory muscles, muscles around the head and neck, ligaments, and teeth. Symptoms seen in temporomandibular dysfunction; pain and tenderness in the muscles and temporomandibular joint; significant or minor limitation of jaw joint movements; clicking sound in the joint during mouth opening and closing, crepitation; a feeling of fullness in the ears, ear pain, tinnitus, and vertigo; emotional disorders such as the deflection of mouth opening, deviation, deterioration in chewing patterns, locking in the jaw, anxiety, depression can be listed as headache. The prevalence of temporomandibular dysfunction in the headache population is 56.1%. It indicates a relationship between temporomandibular dysfunction and headaches' presence, frequency, and intensity. On the other hand, one of the three most common symptoms in temporomandibular dysfunction patients is headache, which is characteristically tension-type. Studies have shown that headache develops in a temporal relationship with temporomandibular disorder and may experience problems such as pain, limitation of movement, and sensitivity. Cognitive changes such as learning, memory, and attention to the painful area that develops with the affected limbic system increase avoidance of movements. However, muscle spasms, pain, negative mood that leads to a vicious circle, and experiences that lead to limitation of movement can be experienced. Therefore, physical and psychosocial factors are also associated with musculoskeletal disorders. The biopsychosocial status of individuals with headaches related to temporomandibular dysfunction should be considered when evaluating treatment efficacy. The pathophysiology of diffuse painful temporomandibular dysfunction is biopsychosocial and multifactorial. Research in this area draws attention to predisposing, initiating, and maintaining factors, including environmental and bodily mechanisms. However, when the literature in this field is examined, it is clear that there is a need for biopsychosocial assessment tools.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 60 years old
* Getting a diagnosis of TMD-related headache
* Not having received FTR and manual therapy in the last 3 months
* Having pain ≥ 50 or more according to the headache impact test (HIT 6)
* Patients who have not received medical treatment in the last 3 months and will not receive medical treatment during the treatment
* Patients who describe pain in the jaw, face, temporal region, or ear for at least 6 months and who have pain in the chewing muscles with palpation

Exclusion Criteria:

* Ages under 18 and over 60 years old
* Patients with disc displacement and attachment degeneration
* Patients with dental infection
* Patients who have undergone facial and ear surgery in the last six months
* Patients undergoing orthodontic treatment
* Patients using regular analgesics or anti-inflammatory drugs
* Patients with a history of trauma (whiplash injury, condylar trauma, fracture),
* Patients who have undergone any surgery related to the cervical and TMJ
* Patients with facial paralysis
* Patients with missing teeth in the upper jaw
* Patients with cognitive deficits
* Participation rate lower than 80% of the program schedule

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with Temporomandibular Dysfunction-Related Headache
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
BETY-Biopsychosocial Questionnaire (BETY-BQ) | 1 week
  The BETY-Biopsychosocial Questionnaire (BETY-BQ) is used to evaluate the biopsychosocial process associated with the disease. A 5-point Likert system is used to score this scale. Each question is scored as "0= never, 1=yes rarely, 2=yes sometimes, 3=yes often, 4=yes always" and gives a total score of over 30 items. A high score means a low biopsychosocial level.

SECONDARY OUTCOMES:
Quality of Life Scale Short Form-36 (SF-36) | 1 week
  Quality of Life Scale Short Form-36 (SF-36) is one of the frequently used scales to measure quality of life. It evaluates eight different categories, such as general health perception, physical function, social function, pain, mental health, role difficulty due to physical reasons, role difficulty due to emotional reasons, and vitality, with a total of 36 sub-items.
  Items are scored as '0 = worst health condition, 100 = best health state'. Each subcategory is scored between 0 and 100 points, with a high score indicating good health.

OTHER OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 1 week
  The Hospital Anxiety and Depression Scale (HADS) is a scale consisting of 14 questions 7 of these questions assess anxiety, and 7 assess depression. Likert-type measurement is used to evaluate this scale. The cut-off score for the anxiety subscale is 10/11, and for the depression, subscale is 7/8. Accordingly, those who score above these scores are considered at risk.
The Jaw Functional Limitation Scale-20 (JFLS-20) | 1 week
  Jaw function limitation will be measured by the Jaw Functional Limitation Scale-20 (JFLS-20), where the patients will be asked for 1 to 10 points per item (higher scores indicate worse jaw function).
  The JFLS-20 has three subscales: Mastication (6 items), Vertical Jaw Mobility (4 items), and Emotional and Verbal Expression (10 items).
The Headache Impact Test (HIT-6) | 1 week
  The Headache Impact Test (HIT-6) consists of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. The patient answers each of the six related questions using one of the following five responses: "never," "rarely," "sometimes," "very often," or "always." These responses are summed to produce a total HIT-6 score that ranges from 36 to 78, where a higher score indicates a greater impact of headaches on the daily life of the respondent. Scores can be interpreted using four groupings that indicate the severity of headache impact on the patient's life.

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur TUNCER, PhD, Study Director — Hasan Kalyoncu University
Locations (1):
- Ayşenur TUNCER, Gaziantep, Hasan Kalyoncu University, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kapos FP, Exposto FG, Oyarzo JF, Durham J. Temporomandibular disorders: a review of current concepts in aetiology, diagnosis and management. Oral Surg. 2020 Nov;13(4):321-334. doi: 10.1111/ors.12473. Epub 2020 Jan 25. PMID 34853604
- [Background] Chisnoiu AM, Picos AM, Popa S, Chisnoiu PD, Lascu L, Picos A, Chisnoiu R. Factors involved in the etiology of temporomandibular disorders - a literature review. Clujul Med. 2015;88(4):473-8. doi: 10.15386/cjmed-485. Epub 2015 Nov 15. PMID 26732121
- [Background] Ohrbach, R., & Sharma, S. (2021). Behavioral therapy for temporomandibular disorders. Frontiers of Oral and Maxillofacial Medicine, 3, 37-37.
- [Background] Oflaz, F.B., Bilişsel Egzersiz Terapi Yaklaşımı Ölçeği'nin Romatoid Artrit Tanısı Alan Bireylerde Geçerliği, Güvenirliği Ve Duyarlılığının Belirlenmesi. 2018, Sağlık Bilimleri Enstitüsü.
- [Background] Kisacik P, Unal E, Akman U, Yapali G, Karabulut E, Akdogan A. Investigating the effects of a multidimensional exercise program on symptoms and antiinflammatory status in female patients with ankylosing spondylitis. Complement Ther Clin Pract. 2016 Feb;22:38-43. doi: 10.1016/j.ctcp.2015.11.002. Epub 2015 Dec 2. PMID 26850804
- [Background] Küçüktepe, İ., et al., Multiple sklerozlu bireylerde Bilişsel Egzersiz Terapi Yaklaşımı'nın yorgunluk ve denge üzerine etkileri. 2018. 5(2): p. 74-81.
- [Background] Edibe, Ü., et al., Romatizmalı hastalar için bir yaşam kalitesi ölçeğinin geliştirilmesi: madde havuzunun oluşturulması. Journal of Exercise Therapy and Rehabilitation 2017. 4(2): p. 67-75.
- [Background] ZAHİD, M., Bilişsel Egzersiz Terapi Yaklaşımı Ölçeği'nin Fibromiyalji Tanısı Alan Bireylerde Geçerliği, Güvenirliği ve Duyarlılığının Belirlenmesi. 2018, Sağlık Bilimleri Enstitüsü
- [Background] Okeson JP. Orofacial pain. In: Guidelines for assessment, diagnosis and management. Chicago: Quintessence Publishing Co;113-184,1996.
- [Background] Günay, Y., Bellaz, İ., Gürgan, C., Gülten, T., & Haskan, H. (1998). Temporomandibular eklem disfonksiyonunda semptomların dağılımı-dıstrubıtıon of semptoms of temporomandıbular joınt dısorder. Journal of Istanbul University Faculty of Dentistry, 32(4), 177-182.
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Skov T, Borg V, Orhede E. Psychosocial and physical risk factors for musculoskeletal disorders of the neck, shoulders, and lower back in salespeople. Occup Environ Med. 1996 May;53(5):351-6. doi: 10.1136/oem.53.5.351. PMID 8673184
- [Background] Ünal, E., Arin, G., Karaca, N. B., Kiraz, S., Akdoğan, A., Kalyoncu, U., ... & Kılıç, L. (2017). Romatizmalı hastalar için bir yaşam kalitesi ölçeğinin geliştirilmesi: madde havuzunun oluşturulması. Journal of Exercise Therapy and Rehabilitation, 4(2): 67-75.
- [Background] Koçyiğit, H., Ö. Aydemir, and G.J.R.h.o.b.g.h.i.ç.İ.v.T.D. Fişek, Kısa Form-36'nın (KF-36) Türkçe için güvenilirliği ve geçerliliği. 1999. 12: p. 102-106.
- [Background] Aydemir, Ö., Güvenir, T., Küey, L., Kültür, S. (1997). Hospital Anxiety and Depression Scale Turkish Form: validation and reliability study. Türk Psikiyatri Der. 8(4): 280-287.
- [Background] https://ubwp.buffalo.edu/rdc-tmdinternational/tmd-assessmentdiagnosis/dc-tmd/dc-tmd-translations
- [Background] Sertel M, Bakar Y, Simsek TT. THE EFFECT OF BODY AWARENESS THERAPY AND AEROBIC EXERCISES ON PAIN AND QUALITY OF LIFE IN THE PATIENTS WITH TENSION TYPE HEADACHE. Afr J Tradit Complement Altern Med. 2017 Jan 13;14(2):288-310. doi: 10.21010/ajtcam.v14i2.31. eCollection 2017. PMID 28573246